CLINICAL TRIAL: NCT04350385
Title: Effects of Dose Response of Plyometric Training on Agility in Cricket Players
Brief Title: Dose Response of Plyometric Training on Agility in Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC/00540 Danish Latif
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Athletic Injuries
Keywords: Agility; Dose Responce; Plyometric training
MeSH Terms: conditions — Athletic Injuries | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Agility Training
  Interventions: Other: Agility training
- Group 2 (Active Comparator): .Conventional intervention
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Agility training — In experimental group, 30 meter sprint test will be used as intervention with complexity in different stages. Test 1 was a straight sprint and tests 2-7 involved multiple changes of direction. Tests 2-7 were designed to involve progressively greater change-of-direction complexity by increasing either the angle of directional change and/or the number of changes of direction. In experimental group, 6 weeks of intervention will be done on alternate days and assessment will be done on 1st, 3rd & 6th week.
  Arms: Group 1
Other: Conventional — In group B, Conventional intervention was given to the players under the supervision of Physical Therapist that includes warm-up, strength training, agility training and cool down. In control group, 6 weeks of intervention will be done on alternate days and assessment will be done on 1st, 3rd & 6th week
  Arms: Group 2

SUMMARY:
The objective of the study was to determine the effects of plyometric training on agility in national cricket players. The study design was Randomized Controlled Trial. 40 cricket players were included in the study through open epi tool out of which n=20 players were in experimental group and n=20 players were in control group. Assessments were taken as baseline on first week, on third week and on sixth week by performing few exercises such as Illinois Agility Run test, T test and Vertical jump test.

DETAILED DESCRIPTION:
Cricket is considered as one of the world's major team sports in terms of regular international games. It is similar to the game of baseball generally played outdoors on natural grass fields. As cricket is a bat and ball sport. Bowling action is explosive in nature; whereby a large amount of force must be generated over a very short period of time. They discussed that fast bowlers have consistently been identified as the category of cricket players at the greatest risk of injury. Bowling action is a highly skilled activity, which is acquired over years of fine tuning. Equally from a neuromuscular perspective, the bowling action is a complex activity and optimal performance is a result of highly tuned inter-muscular and intra-muscular coordination, which is governed by the central nervous system. It has been shown that recently modern training techniques and in particularly strength training, has been perceived to be a major contributing factor to the recent injuries sustained at a national level.

In many sports straight sprinting speed and agility are considered important qualities. Straight line sprinting is a relatively closed skill involving predictable and planned movements and is used in sports such as track and field and gymnastics. It is difficult to define agility, as it is the ability to change direction and start and stop quickly. In a sporting situation, changes of direction may be initiated to either pursue or evade an opponent or react to a moving ball. Therefore, it has been recognized that a component of agility performance is the response to a stimulus. Further Chelladurai and Yuhasz demonstrated that a change of direction task with a simple stimulus shared only 31% common variance with a more complex task in which the timing and location of the stimulus were not known. It has been shown that up-and-back sprint time of 2.4-m increased as a light stimulus became less predictable in terms of timing and location, presumably because of increased information processing.This suggests that having to react to a stimulus such as an opponent's movement on the field may significantly influence the nature of the change-of-direction movement task.

Several studies have reported correlations between straight sprint tests and various agility tests. When a correlation coefficient (r) is less than 0.71, the shared or common variance between the 2 variables is less than 50%, indicating that they are specific or somewhat independent in nature. Hortobagyi et al. used this statistical approach to demonstrate that various modes of strength testing indicated more generality (r ˃ 0.71) of strength than specificity (r ˂ 0.71). Common variances of 11% and 22% have been reported, respectively, for straight sprints and a soccer agility test and the Illinois agility test. Further, these investigators conducted a factor analysis on several fitness test results and found the speed and agility tests to be represented by different factors. This meant that speed and agility had little in common statistically, leading the authors to conclude that they were relatively independent qualities.

In 1969, a study was conducted that compared the effects of speed and agility training on various fitness parameters. The study reported that agility training was superior to speed training for performance in the Illinois agility run and a ''zig-zag run'' but the speed training was not significantly better for improving 50-yd sprint time. Unfortunately, the authors failed to describe the training that was implemented, making it difficult to evaluate the effects. Since the potential specificity of speed and agility training has not yet been clearly established, the purpose of the present study was to determine if straight sprint training transferred to change-of-direction tests of varying complexities. Another objective was to determine if agility training could enhance straight sprinting speed. Plyometric consists of a rapid stretching of a muscle (eccentric action) immediately followed by a concentric or shortening action of the same muscle and connective tissue. Plyometric drills usually involve stopping, starting, and changing directions in an explosive manner. These movements are components that can assist in developing agility. Plyometric exercises include jumps, hops, skips, bounds and throws. Plyometric training is an intense form of exercise that helps athletes improves the power of their movements. Plyometric training is used to improve maximum strength and speed of movement which result in an increase of explosive power.

Agility is the ability to change direction or body position rapidly and proceed with another movement. Agility is the physical ability that enables a person rapidly to change body position and direction in a precise manner. Agility is generally defined as the ability to change direction quickly and effectively while moving as possible at full speed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-25 Years.
* Males
* Those who had minimum one year of experience in domestic cricket(first class)

Exclusion Criteria:

- Players undergone surgery or had accident within last 6 months.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Agility T test | 6th week
  In T test players have to run 40 yards and time will be noted in seconds. Rating starts from >11.5 seconds (poor) to <9.5 seconds (excellent).
Illinios agility test | 6th week
  Player have to run about 60 meters and time will be noted in seconds with rating poor >18.8 seconds and excellent <15.9 seconds.
vertical jump height | 6th week
  The testing subject stood on side of wall and reached her hand at it max. The foot was kept flat on the ground. The finger tip of hand was marked as standing normal max. Distance with foot flat. This was recorded as standing reach height.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, *PHD, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rae K, Orchard J. The Orchard Sports Injury Classification System (OSICS) version 10. Clin J Sport Med. 2007 May;17(3):201-4. doi: 10.1097/JSM.0b013e318059b536. PMID 17513912
- [Background] Karppinen S, editor Strength training for fast bowlers: Resistance to resistance training. 1 of 1-Conference of Science, Medicine & Coaching in Cricket 2010; 2010
- [Background] Young WB, McDowell MH, Scarlett BJ. Specificity of sprint and agility training methods. J Strength Cond Res. 2001 Aug;15(3):315-9. PMID 11710657
- [Background] Chelladurai P. Manifestations of agility. Journal of the Canadian Association of Health, Physical Education and Recreation. 1976;42(3):36-41.
- [Background] Chelladurai P, Yuhasz M, Sipura R. The reactive agility test. Perceptual and Motor Skills. 1977;44(3_suppl):1319-24.
- [Background] Thomas JR, Silverman S, Nelson J. Research methods in physical activity, 7E: Human kinetics; 2015.
- [Background] Hortobagyi T, Katch FI, LaChance PF. Interrelationships among various measures of upper body strength assessed by different contraction modes. Evidence for a general strength component. Eur J Appl Physiol Occup Physiol. 1989;58(7):749-55. doi: 10.1007/BF00637387. PMID 2737196
- [Background] Buttifant D, Graham K, Cross K, editors. Agility and speed measurement in soccer players are two different performance parameters. Fourth World Congress of Science and Football; 1999.
- [Background] Draper J. The 505 test: A test for agility in horizontal plane. Aust J Sci Med Sport. 1985;17(1):15-8.
- [Background] Mayhew J, Piper F, Schwegler T, Ball T. Contributions of speed, agility and body composition to anaerobic power measurement in college football players. The Journal of Strength & Conditioning Research. 1989;3(4):101-6.
- [Background] Hilsendager DR, Strow MH, Ackerman KJ. Comparison of speed, stength, and agility exercises in the development of agility. Res Q. 1969 Mar;40(1):71-5. No abstract available. PMID 5252467
- [Background] Craig BW. What is the scientific basis of speed and agility? Strength & Conditioning Journal. 2004;26(3):13-4.
- [Background] Gabbard C, LeBlanc E, Lowy S. Physical education for children: Building the foundation: Prentice-Hall; 1994
- [Background] Singer RN. Motor learning and human performance: An application to physical education skills: Macmillan; 1975.